CLINICAL TRIAL: NCT05189067
Title: A Single-center, Prospective, Randomized Study of Adjuvant Paclitaxel and Trastuzumab Versus Docetaxel and Trastuzumab in Stage I HER2 Positive Breast Cancer
Brief Title: Efficacy and Safety of Adjuvant Docetaxel and Trastuzumab in Stage I HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0170
Record Dates: First submitted 2021-12-06; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-11

CONDITIONS: HER2-positive Breast Cancer; Adjuvant Therapy
Keywords: Docetaxel; Paclitaxel
MeSH Terms: interventions — Paclitaxel; Trastuzumab; Protons; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paclitaxel + trastuzumab (Active Comparator): paclitaxel × 12, every week a cycle, trastuzumab × 4, every 3 weeks a cycle; followed by trastuzumab, every 3 weeks a cycle for 9 months.
  Paclitaxel i.v. 80mg/m2, trastuzumab i.v. loading dose of 8 mg/kg, followed by 6mg/kg
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab
- docetaxel + trastuzumab (Experimental): (docetaxel + trastuzumab) × 4, every 3 weeks a cycle; followed by trastuzumab, every 3 weeks a cycle for 9 months.
  Docetaxel i.v. 100mg/m2, trastuzumab i.v. loading dose of 8 mg/kg, followed by 6mg/kg
  Interventions: Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Paclitaxel — i.v. 80mg/m^2
  Other Names: P
  Arms: paclitaxel + trastuzumab
Drug: Trastuzumab — i.v. loading dose of 8 mg/kg, followed by 6mg/kg
  Other Names: H
Drug: Docetaxel — i.v. 100mg/m2
  Other Names: T
  Arms: docetaxel + trastuzumab

SUMMARY:
Among women with stage I HER2-positive breast cancer, adjuvant weekly paclitaxel plus trastuzumab (PH, qw×12) is one of the standard therapies. However, it is quite inconvenient for patients to received weekly treatment for 12 weeks, which also increased the patients' and social economic burdens. In our study, a prospective, randomized, open-label, single-center clinical study was conducted to compare the efficacy and safety of adjuvant docetaxel plus trastuzumab (TH, q3w×4) and the classic regimen (PH, qw×12) in stage I HER2-positive breast cancer in Chinese population.

DETAILED DESCRIPTION:
HER2-positive breast cancer accounts for about 20% of invasive breast cancers and was historically associated with poor clinical outcomes. Trastuzumab, a humanized monoclonal antibody that binds HER2, improved the outcomes for patients with HER2-positive breast cancer. Four phase 3 randomized trials (HERA, the North Central Cancer Treatment Group N9831, the National Surgical Adjuvant Breast and Bowel Project B-31 and BCIRG006) involving more than 8000 patients showed that when trastuzumab was administered in combination with or after chemotherapy, the risk of recurrence was decreased by approximately 50% and overall survival improved.

For patients with lymph node negative, early stage HER2-positive breast cancer, epirubicin/cyclophosphamide followed by docetaxel/trastuzumab (AC-TH) or docetaxel/carboplatin/trastuzumab (TCbH) adjuvant regimen is still widely used, although a smaller absolute benefit is expected. According to the long-term survival outcome of the Adjuvant Paclitaxel and Trastuzumab (APT) trial, patients with tumors measuring up to 3 cm in greatest dimension, negative axillary lymph node or with only micrometastasis, who received adjuvant paclitaxel 80mg/m2 weekly for 12 times plus 1 year trastuzumab, achieved a 3-year disease free survival (DFS) of 98.5%, 5-year DFS of 96.3%, 7-year DFS of 93.3%. The FDA compared the outcome of APT trial with external controls from previous clinical trials, both DFS and overall survival (OS) were similar.

However, weekly regimen is quite inconvenient for patients, which also increased the patients'and social economic burdens in China. Docetaxel, a newly developed taxoid anticancer agent, works a comparable way to paclitaxel. In the clinical trial E1199, early breast cancer patients receiving adjuvant adriamycin and cyclophosphamide (AC) followed by docetaxel every 3 weeks achieved similar outcomes with AC followed weekly paclitaxel. In our study, a prospective, randomized, open-label, single-center clinical study is conducted to compare the efficacy and safety of adjuvant docetaxel plus trastuzumab (TH, q3w×4) and the classic regimen (PH, qw×12) in stage I HER2-positive breast cancer in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 - 70 years old;
2. The histopathological confirm of invasive breast cancer;
3. HER-2 positive: immuno-histochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) confirmed amplification of erbb2 gene;
4. Tumor must be ≤ 2cm in greatest dimension, negative axillary lymph node or with micrometastasis (axillary nodes with tumor clusters ≤ 0.2cm);
5. No more than 90 days from the patient's most recent breast surgery for this breast cancer;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
7. Adequate bone marrow function: neutrophil ≥ 1500/mm^3, hemoglobin ≥ 9 g/dl, and platelets ≥ 100,000/mm^3;
8. Adequate liver and renal function: creatinine ≤ 1.5 folds of the upper limit of normal value; aspartate aminotransferase and alanine aminotransferase ≤ 1.5 folds of the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2 folds of the upper limit of normal value for patient with Gilbert 's syndrome;
9. Left ventricular ejection fraction (LVEF) ≥ 50%;
10. Willing and able to sign informed consent.

Exclusion Criteria:

1. Any of the following due to teratogenic potential of chemotherapy: pregnant women, nursing women, women of childbearing potential who are unwilling to employ adequate contraception;
2. Locally advanced tumors at diagnosis, including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes;
3. History of prior chemotherapy in the past 5 years;
4. History of prior trastuzumab therapy;
5. Patients with a history of previous invasive breast cancer;
6. Active, unresolved infection;
7. Prior history of any other malignancy in the past 5 years, except for early stage tumors of the skin or cervix treated with curative intent;
8. Can not tolerate or be allergic to chemotherapy, anti-HER-2 therapy or pharmaceutical materials such as benzyl alcohol;
9. ≥ grade 2 neuropathy;
10. Active cardiac disease: Any prior myocardial infarction (asymptomatic changes on EKG suggestive of old myocardial infarction is not an exclusion); Documented congestive heart failure (CHF); Current use of any therapy specifically for CHF; Current uncontrolled hypertension (diastolic >100 mmHg or systolic > 200 mmHg); Clinically significant pericardial effusion;
11. The antibody of hepatitis C virus, HIV or Treponema pallidum positive; HBsAg positive and hepatitis B virus DNA in peripheral blood ≥ 10^3 copy/mL；
12. Enrollment on other Investigational studies within 30 days;
13. Not allowed by the investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | Time of Surgery up to 5 years
  Evaluate disease free survival (DFS) in patients with stage I HER2-positive breast cancer treated with adjuvant trastuzumab and docetaxel.

SECONDARY OUTCOMES:
overall survival | Time of Surgery up to 5 years
  Evaluate overall survival (OS) in patients with stage I HER2-positive breast cancer treated with adjuvant trastuzumab and docetaxel.
incidence of grade III/IV neurotoxicity | First Dose of chemotherapy up to 12 months.
  Evaluate the incidence of grade III/IV neurotoxicity associated with adjuvant docetaxel compared with paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Pan, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No